CLINICAL TRIAL: NCT00633087
Title: A Phase I/II Trial of 2-Deoxyglucose (2DG) for the Treatment of Advanced Cancer and Hormone Refractory Prostate Cancer
Acronym: 2-Deoxyglucose
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080402; IRB# 0220044763 (Other: IRB)
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Deoxyglucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2-deoxyglucose (Experimental)
  Interventions: Drug: 2-deoxyglucose

INTERVENTIONS:
Drug: 2-deoxyglucose — 30 mg/kg of 2-deoxyglucose administered orally on a daily schedule for two weeks (Days 1-14) of a three week (21 Day) cycle.
  Other Names: Two-deoxyglucose

SUMMARY:
Subjects will be asked to participate in this clinical trial to examine the safety of 2-deoxyglucose (an agent which is quite similar to glucose) in the treatment of solid tumors and hormone refractory prostate cancer. This agent works by blocking the metabolism of glucose in the cells of the body. Although all cells require glucose for metabolism, it is believed that cancer cells require significantly more glucose than normal cells to grow. Therefore, even slight effects of glucose metabolism in cancer cells might result in the shrinkage of certain cancers. This agent has been given to humans before and has only caused mild nausea, vomiting and glucopenia (low blood sugar) at the doses given in these studies. This study will further examine the safety of 2-deoxyglucose in the treatment of advanced solid tumors and hormone refractory prostate cancer. The information obtained in this study will be used to design future clinical studies with 2-deoxyglucose. Subjects will be asked to take an oral solution of 2-deoxyglucose daily, by mouth, while on this study. They will be asked to have CT Scans, Bone Scans, and optional PET (Positron Emission Tomography) Scans prior to starting this study. PET scans will also be performed shortly after the start of the study and after 2 cycles (6 weeks) of therapy. Subjects will be asked to have a comprehensive physical examination and blood work prior to the start of the study. During the first 2 cycles of the study subjects will be asked to have blood drawn at different time intervals for the first 2 days of each cycle. While on the study, they will be asked to return to the clinic at intervals of 1 week for a physical examination and blood tests. Subjects will also be asked to have CT Scans and Bone Scans at intervals of 9 weeks while on the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any histologically proven metastatic solid tumor malignancy, without a standard option of therapy will be eligible for the Phase I portion of this trial. Patients with prostate cancer with metastatic disease, and progression after initial hormonal therapy will be eligible for both the Phase I and II portion of this trial. Phase II patients must have either measurable disease or a PSA value > 5 ng/ml.
* Patients with prostate cancer in whom bicalutamide or flutamide has been recently withdrawn, must demonstrate progression of disease and be at least 6 weeks and 4 weeks respectively beyond the discontinuation of such agents. LHRH agonists will be continued.
* Age >18 years and an estimated life expectancy of at least 6 months.
* ECOG performance status < 2. (see Appendix B)
* Patients must be ³ 4 weeks since last prior therapy (including surgery, chemotherapy, radiation therapy). All previous clinically significant treatment-related toxicities have resolved to less than or equal to Grade 1.
* An ANC >1500/µl, hemoglobin > 10 g/dl, and platelet count >100,000/µl are required.
* Adequate renal function (serum creatinine < 1.5 mg/dL or creatinine clearance > 50 ml/min)
* Total bilirubin must be within normal limits. Transaminases (SGOT and/or SGPT) must be less than 2.5X the institutional upper limit of normal.
* Serum potassium within institutional limit of normal.
* Fasting blood glucose < institutional ULN.
* In the Phase I portion of this study patients may have had prior chemotherapy.
* In the Phase II portion of this study patients may not have had prior chemotherapy.
* Women of childbearing potential must have a negative pregnancy test (Phase I trial).
* Men and women of childbearing potential must consent to using effective contraception while on treatment and for 3 months thereafter.

Exclusion Criteria:

* Known infection with HIV. Patients without prior HIV testing will not be required to be tested.
* History of glucose intolerance.
* Patients with ongoing coagulopathies and/or receiving oral anticoagulants.
* Second primary malignancy except most situ carcinoma (e.g. in situ carcinoma of the of the cervix, adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least 5 years previously with no evidence of recurrence.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with diabetes mellitus, hypoglycemia, history of seizure disorder, known autonomic dysfunction, clinically significant uncontrolled gastrointestinal disorder, known G6PD deficiency, and allergy to methylparaben or propylparaben will be excluded, based on known potential toxicities.
* The effects of 2-deoxyglucose on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because Agent Class as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 3 months thereafter. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Active clinically significant infection requiring antibiotics.
* History of clinically significant unexplained episodes of hypotension, fainting, dizziness, or lightheadedness.5.2.10 History or symptoms of cardiovascular disease (NYHA Class 2, 3, or 4; see Appendix D, New York Heart Association Criteria) within the last 6 months, particularly coronary artery disease, arrhythmias, or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, or congestive heart failure.
* History of transient ischemic attack, stroke, or seizure disorder or any other CNS disease considered to be significant by the investigator.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Antitumor therapy within 28 days of the start of study treatment (within 6 or 4 weeks for bicalutamide or flutamide, respectively).
* Phase I only: Inability to discontinue prohibited medications for 24 hours before and after dosing on Cycle 1, Day 1 of Weeks 1 and 2.
* Patients who are unable (as per Investigator discretion) or unwilling to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert DiPaola, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- The Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve subjects were enrolled from April 2007 through June 2009 at The Cancer Institute of New Jersey, a comprehensive cancer center.
Groups:
- 2-deoxyglucose: 2-deoxyglucose : 30 mg/kg of 2-deoxyglucose administered orally on a daily schedule for two weeks (Days 1-14) of a three week (21 Day) cycle.
Period: Overall Study
Arm/Group | 2-deoxyglucose
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 2-deoxyglucose
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Biochemical Response of This Regimen in Patients With HRPC
Description: A PSA response is defined as a PSA decrease of 50% from baseline maintained for at least 28 days.
Time Frame: 5 years
Population: No data collected
Arm/Group | 2-deoxyglucose
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Time Frame: 5 years
Population: No data collected
Arm/Group | 2-deoxyglucose
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | 2-deoxyglucose
Number analyzed (Participants) | 12
Participants | 9

4. Secondary Outcome: Overall Survival
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | 2-deoxyglucose
Number analyzed (Participants) | 12
Participants | 7

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | 2-deoxyglucose
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-deoxyglucose (N=12)
Pain - Back (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Pain (right lower quadrant) (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-deoxyglucose (N=12)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (8)
Prolonged QTc interval (Cardiac disorders) | 4 (4)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 1 (3)
Pain (General disorders) | 2 (2)
Pain - Back (General disorders) | 1 (2)
Pain - Chest wall (General disorders) | 1 (1)
Pain - Pelvis (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (nose) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes